CLINICAL TRIAL: NCT06233656
Title: Acceptance and Commitment Therapy for Depressed People With Spinal Cord Injuries: Testing Efficacy and Mechanisms of Change
Brief Title: Acceptance and Commitment Therapy for Depressed People With Spinal Cord Injuries
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Areum Han, Associate Professor, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300012385; 1077500 (Other Grant/Funding Number: Craig H. Neilsen Foundation)
Record Dates: First submitted 2024-01-15; First posted 2024-01-31 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Depression; Spinal Cord Injuries
Keywords: Acceptance and Commitment Therapy; Depression; Mindfulness; Spinal cord injuries
MeSH Terms: conditions — Depression; Spinal Cord Injuries | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and commitment therapy (ACT) group (Experimental): The ACT group will receive eight weekly individual ACT sessions guided by a coach through videoconferencing with a booster session at 1-month follow-up.
  Interventions: Behavioral: Acceptance and commitment therapy (ACT)
- Wait-list control group (No Intervention): The wait-list control group will maintain his or her own care as usual during the study period and receive eight individual ACT sessions after study participation ends.

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy (ACT) — Participants assigned to the ACT group will receive 8 weekly individual ACT sessions guided by a coach for one hour per week over 8 weeks through Zoom videoconferencing.
  Arms: Acceptance and commitment therapy (ACT) group

SUMMARY:
Living with spinal cord injury (SCI) can have a significant negative impact on an individual's mental health and restrict participation in personally valued activities and roles. Acceptance and commitment therapy (ACT) is an evidence-based approach that can lessen symptoms of mental health disorders (e.g., depressive symptoms) and improve quality of life through mindfulness and acceptance processes and behavior change processes for valued living. Evidence for ACT for individuals living with SCI, however, is limited to a very few studies that involved in-person group-based ACT and did not focus on depressed individuals with SCI.

The primary goal of this study is to evaluate the effects of an 8-week videoconferencing ACT program on improving mental health outcomes in depressed individuals living with SCI. The primary hypotheses are that the ACT group will show improvements in depressive symptoms at posttest and 2-month follow-up compared to the wait-list control group. Investigators will invite 120 individuals living with SCI and reporting depressive symptoms and randomly assign them to either the ACT group or the wait-list control group. The ACT group will receive eight weekly individual ACT sessions guided by a coach through videoconferencing with a booster session at 1-month follow-up. The wait-list control group will continue his or her own care as usual during the study period and have the option to receive eight individual ACT sessions after study participation ends. Data will be collected at pretest, posttest, and 2-month follow-up and compared between the ACT group and the control group over time.

About 40% of individuals living with SCI report depressive symptoms and other mental health symptoms, and mental health disorders following SCI are associated with negative long-term outcomes. Managing uncomfortable or painful thoughts and emotions arising from functional limitations and accepting changed lives while moving forward for valued living through ACT skill practice will help individuals with SCI alleviate symptoms of mental health conditions, promote engagement in personally valued activities, and improve quality of life.

DETAILED DESCRIPTION:
Living with spinal cord injury (SCI) can have a significant negative impact on an individual's mental health and restrict participation in personally valued activities and roles. About 40% of individuals with SCI report depressive symptoms and other mental health symptoms, which are associated with negative long-term outcomes.

Acceptance and commitment therapy (ACT) is an empirically supported transdiagnostic approach that can mitigate symptoms of mental health disorders and improve quality of life through mindfulness and acceptance processes and behavior change processes for valued living. ACT is based on the psychological flexibility model involving six processes that serve as a mechanism of change (i.e., acceptance, cognitive defusion, being present, observing self, values, and committed action). Evidence for ACT for individuals with SCI, however, is limited to a very few studies that involved in-person group-based ACT and did not focus on depressed individuals with SCI.

This project aims to test the efficacy of an 8-week videoconferencing ACT program for improving mental health in depressed individuals living with SCI. The hypotheses are that the ACT group will show improvements in depressive symptoms (the primary outcome), secondary mental health outcomes (e.g., anxiety, stress, and grief), and ACT processes (e.g., psychological flexibility and engaged living) at posttest and 2-month follow-up compared to the wait-list control group. Also, the project aims to examine the mediating effects of the ACT psychological flexibility processes on reducing depressive symptoms in individuals living with SCI.

This study will use a two-arm parallel-group, randomized controlled trial design. The investigators will recruit approximately 120-140 depressed individuals living with SCI and randomly assign them to either the ACT group or the wait-list control group. The ACT group will receive eight weekly individual ACT sessions guided by a coach through videoconferencing with a booster session at 1-month follow-up. The wait-list control group will maintain his or her own care as usual during the study period and have the option to receive eight individual ACT sessions after study participation ends. Data will be collected at pretest, posttest, and 2-month follow-up. The investigators will use generalized linear mixed-effects models to examine the relative impact on the ACT group compared to the wait-list control group at posttest and 2-month follow-up. The mediation analysis will consist of the outcome model and the mediator model. After fitting the models, the investigators will estimate direct effect and indirect effect (i.e., the mediated effect).

Managing uncomfortable or painful thoughts and emotions arising from functional limitations and accepting changed lives while moving forward for valued living through ACT skill practice will help individuals with SCI alleviate symptoms of mental health conditions, promote engagement in personally valued activities, and improve quality of life. The investigators expect the findings of this study to contribute to the limited evidence for internet-delivered ACT in individuals living with SCI and lay the necessary groundwork to provide important knowledge and guidance for future clinical trials and practice.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling adults (aged 18 years or older) living with spinal cord injuries
* having at least mild depressive symptoms as measured by the PHQ-9 (scores ≥ 5)
* having a web-enabled device (e.g., a computer or a smartphone) with internet access

Exclusion Criteria:

* having cognitive deficits or language barriers that might impede study participation
* having suicidal intent or attempts in the past 6 months
* having psychiatric hospitalizations in the previous 2 years
* having a diagnosis with bipolar disorder or psychotic disorders (e.g., schizophrenia)
* having a prior experience with acceptance and commitment therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up on the Patient Health Questionnaire-9 (PHQ-9) | Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up
  The PHQ-9 is a 9-item questionnaire assessing depressive symptoms on a scale of 0 to 3. Scores range from 0 to 27. Higher scores indicate greater symptomatology in depression.

SECONDARY OUTCOMES:
Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up on the Spinal Cord Injury-Quality of Life (SCI-QOL) Depression Short form | Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up
  The SCI-QOL Depression Short form (a back-up measure of depressive symptoms) has 10 items assessing the severity of depressive symptoms in individuals living with SCI on a scale of 1 (never) to 5 (always). Scores range from 10 to 50, and higher scores indicate higher levels of depressive symptoms.
Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up on the Generalized Anxiety Disorder-7 (GAD-7) | Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up
  The GAD-7 is a 7-item questionnaire assessing anxiety on a scale of 0 to 3. Scores range from 0 to 21. Higher scores indicate greater anxiety.
Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up on the Perceived Stress Scale - 10 (PSS-10) | Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up
  The PSS-10 is a 10-item questionnaire assessing stress on a scale of 0 to 4. Scores range from 0 to 40. Higher scores indicate greater stress
Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up on the World Health Organization Quality of Life (WHOQOL) - Psychological health component | Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up
  The WHOQOL - Psychological health component has 6 items measuring psychological quality of life on scale of 1 to 5. Scores range from 6 to 30. Higher scores denote higher quality of life in terms of psychological health.
Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up on the Spinal Cord Injury-Quality of Life (SCI-QOL) Grief and Loss Short form | Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up
  The SCI-QOL Grief and Loss Short form has nine items assessing grief and loss due to SCI on a scale of 1 to 5. Scores range from 9 to 45, and higher scores indicate more grief and loss.
Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up on the SCI-QOL Resilience Short form | Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up
  The SCI-QOL Resilience Short form has eight items assessing resilience on a scale of 1 to 5. Scores range from 8 to 40, and higher scores indicate greater resilience.
Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up on the Self-Compassion Scale - Short Form (SCS-SF) | Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up
  The SCS-SF is a 12-item self-report questionnaire assessing self-compassion on a scale of 1 to 5. Scores range from 12 to 60. Higher scores indicate higher levels of self-compassion.
Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up on the Multidimensional Psychological Flexibility Inventory - 24 (MPFI-24) | Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up
  The MPFI-24 is a 24-item self-report questionnaire measuring psychological flexibility /inflexibility on a scale of 1 to 6. Scores on pairs of items are averaged to represent each of the 12 specific dimensions of psychological flexibility and inflexibility. The averages of the 6 flexibility subscales can be averaged to create a composite representing global flexibility (i.e., higher scores indicates greater psychological flexibility). Similarly, the averages of the 6 inflexibility subscales can be averaged to create a global inflexibility composite (i.e., higher scores indicate greater psychological inflexibility).
Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up on the Action and Acceptance Questionnaire-II (AAQ-II) | Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up
  The AAQ-II is a 7-item self-report questionnaire measuring experiential avoidance on a scale of 1 to 7. Scores range from 7 to 49. Higher scores indicate greater experiential avoidance.
Change from baseline to immediately after the intervention (or 2 weeks) and 2 month follow-up on the Cognitive Fusion Questionnaire -7 (CFQ-7) | Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up
  The CFQ-7 is a 7-item self-report questionnaire measuring cognitive fusion on scale of 1 to 7. Scores range from 7 to 49. Higher scores indicate greater levels of cognitive fusion.
Change from baseline to immediately after the intervention (or 8 weeks) and 2-month follow-up on the Engaged Living Scale -9 (ELS-9) | Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up
  The ELS-9 is a 9-item self-assessment instrument that measures clarity and engagement with personal values on a scale of 1 to 5. The total scores range from 9 to 45, and higher scores indicate increased clarity and engagement with personal values.
Change from baseline to immediately after the intervention (or 8 weeks) and 2-month follow-up on the Five Facet Mindfulness Questionnaire - Short Form (FFMQ-SF) | Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up
  The FFMQ-SF is a 24-item questionnaire assessing five facets of mindfulness (i.e., observing, describing, acting with awareness, non-judgment of inner experiences, and non-reactivity to inner experiences) on a scale of 1 (never or very rarely true) to 5 (very often or always true). Facet scores range from 5 to 25 (except for the observing facet, which ranges from 4 to 20), and higher scores reflect higher levels of mindfulness.
Change from baseline to immediately after the intervention (or 8 weeks) and 2-month follow-up on the Satisfaction with Life Scale (SWLS) | Change from baseline to immediately after the intervention (or 8 weeks) and 2 month follow-up
  The SWLS is a short 5-item questionnaire assessing satisfaction with one's life on a scale of 1 (Strongly disagree) to 7 (Strongly agree). Scores range from 5 to 35 and higher scores reflect higher life satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Areum Han, PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No